CLINICAL TRIAL: NCT00407368
Title: Platelets Function and Cardiovascular Events in Patients With End Stage Renal Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 75/06
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-11

CONDITIONS: End Stage Renal Disease; Cardiovascular Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood Sample

SUMMARY:
The purpose of this study is to perform a prospective evaluation regarding the relationship between platelets function and cardiovascular events in patients with ESRD.

The study will include 100-200 patients with ESRD, age 18 years or older, treated in the nephrology division of Assaf Harofeh medical center.

The primary end points of the study are cardiovascular events including acute myocardial infarction (defined as symptoms + acute elevation of TnI), need for coronary artery disease revascularization, or acute cerebrovascular event (TIA or CVA) and mortality. The secondary end points are any hospitalization due to acute coronary syndrome, active bleeding with the need for blood transfusion and dialysis access graft thrombosis (time to thrombosis).

Blood will be taken for complete blood count including platelets count and mean platelets volume, serum electrolytes, albumin, blood lipids, Kt/V, troponin and two 5 ml aliquots from each blood collection will be separated and stored at -70co until analyzed for oxidative stress, homocysteine and highly sensitive CRP will be performed. Five mL of blood will be sent for platelets function assessment.

During the follow up period the correlation between platelets function an cardiovascular events will be assessed.

DETAILED DESCRIPTION:
Background Platelets play an important role in cardiovascular disease both in the pathogenesis of atherosclerosis and in the development of acute thrombotic events. Their importance in coronary disease and in acute coronary syndromes is indirectly confirmed by the benefit of antiplatelet agents (particularly aspirin, clopidogrel, ticlopidine, and the glycoprotein IIb/IIIa inhibitors) in these disorders. Cardiovascular disease is the single best predictor of mortality in patients with end-stage renal disease, as it accounts for almost 50 percent of deaths. Patients with end stage renal disease (ESRD) have an increased tendency to bleeding due to platelet dysfunction that can be partly corrected by either hemodialysis or peritoneal dialysis in approximately two-thirds of cases. Currently there is only scant data concerning the relations between platelet function and cardiovascular risk in patients with ESRD.

Platelets, platelet products, and thrombosis play important and proximate causal roles in the occurrence of acute occlusive vascular events such as MI and ischemic stroke. The disruption of platelet and fibrin rich atherosclerotic plaques may lead to enhanced platelet deposition, and ultimately the formation of a thrombus that can precipitate an acute clinical event. The following observations are compatible with the importance of platelet thrombus formation in acute ischemic syndromes:

* Thrombus formation within a coronary vessel is the acute precipitating event in most unstable ischemic coronary syndromes, as documented by angiographic and pathologic studies . Among patients with sudden death due to coronary thrombosis, the thrombi typically have a layered appearance indicative of episodic growth. Episodic growth may alternate with intermittent fragmentation of the thrombus, leading to distal embolization of both thrombus and platelet aggregates and microinfarction.
* Increased platelet-derived thromboxane A2 and other prostaglandin metabolites have been found in patients with acute myocardial infarction and unstable angina, providing biochemical support for platelet activation as the cause of these events.
* Patients with unstable angina have elevated levels of P-selectin, an integral membrane protein involved in platelet adhesion. Pulsatile shear stress, as occurs in stenotic arteries, can cause platelet aggregation via an increased expression of P-selectin. Hydrodynamic shear stress, resulting from plaque rupture, can activate platelets and cause both platelet aggregation (via glycoprotein IIb/IIIa and von Willebrand factor) and platelet-mediated neutrophil aggregation via upregulation of P-selectin. Although levels of P-selectin decrease during the first month after treatment, levels remain higher than normal even with therapy with glycoprotein IIb/IIIa inhibitors, suggesting continued platelet activation.
* Aggregating platelets from patients with acute coronary syndromes produce less nitric oxide than those from patients with stable or no angina. Why this might occur is not known, but impaired nitric oxide production can enhance platelet aggregation and thrombus formation.

Another platelet-related factor believed to contribute to cardiovascular thrombosis is the presence of larger, more reactive platelets in patients with acute ischemic events (19-21). The increase in platelet size, which is in compensation for a persistent decrease in platelet count, results from the ongoing consumption of platelets in unstable angina; this is not seen in an acute myocardial infarction. In addition, platelets from patients with unstable angina, as determined by studying platelet aggregability ex vivo, are hyperaggregable. These effects promote thrombus growth, limitation of blood flow, and acute ischemia.

Except for the important of platelets in occlusive vascular events several studies suggests that they may also have a role in the evolutionary phase of the atherosclerotic plaque. After adhesion to exposed subendothelium following endothelial injury they release vasoactive substances that induce smooth muscle cell migration and proliferation. Platelets may serve as a lipid source in the development of the fatty streak and can promote foam cell formation even in the absence of hyperlipidemia. However, currently there is no clear clinical evidence that platelets contribute to coronary atherosclerosis. In addition, prophylactic therapy with aspirin has not been clearly shown to decrease the atherosclerotic burden.

ESRD is associated with prolongation of the bleeding time due primarily impaired platelet function. It is likely that multiple factors are responsible for the platelet dysfunction in uremia. Three of the factors that may contribute are the retention of uremic toxins, anemia, and nitric oxide.

* Uremic toxins - The importance of circulating toxins is suggested by the often beneficial effect of acute dialysis on platelet dysfunction, although the bleeding time is rarely normalized. In addition, raising the BUN to 60 to 120 mg/dL by dietary manipulation can diminish platelet adhesiveness and prolong the bleeding time in some normal subjects. Urea alone, however, is probably not the major platelet toxin and there is no predictable correlation between the BUN and the bleeding time in patients with renal failure. Other potential toxins include guanidinosuccinic acid, phenolic acid, and middle molecules (mol wt 500 to 3000 daltons). In vitro studies in which normal platelets are incubated with uremic serum suggest that a dialyzable factor interferes with the binding of fibrinogen to the platelet glycoprotein (GP) IIb/IIIa receptor. In addition, uremic platelets are unable to adequately increase the expression of GP IIb/IIIa and P-selectin in response to stimulation.
* Anemia - Previously, anemia was a common finding in chronic renal failure. The degree of anemia appears to correlate relatively closely with the degree of prolongation of the bleeding time. Furthermore, correction of anemia with blood transfusions or erythropoietin often improves platelet function. It has been proposed that the rheologic factors play an important role in the relationship between anemia and platelet dysfunction. At a hematocrit above 30 percent, the red cells primarily occupy the center of the vessel, while the platelets are in a skimming layer at the endothelial surface. This close proximity allows the platelets to adhere and then form a platelet plug when there is endothelial injury. With anemia, on the other hand, the platelets are more dispersed, thereby impairing adherence to the endothelium.
* Nitric oxide - Nitric oxide (NO; endothelium-derived relaxing factor) is an inhibitor of platelet aggregation that is produced by endothelial cells and platelets. Studies in uremic patients have shown that platelet NO synthesis is increased and that uremic plasma stimulates NO production by cultured endothelial cells. The increase in NO synthesis may be due to elevated levels of guanidinosuccinic acid, a uremic toxin that may be a precursor for nitric oxide in this setting.

Although patients with ESRD are at increase risk for cardiovascular disease there are only scant data concerning the cardioprotective effect of antiplatelets drugs for primary or secondary prevention in this population. In a retrospective evaluation of patients with ESRD after acute myocardial infarction, Berger et al. have found that aspirin is underused in this population (67.0%) and Similar results were found by McCullough et al., . Balanced against the potential, but unproven benefit of aspirin in patients with ESRD are its potential risks, including bleeding and a possible acceleration of access thrombosis. The evidence for accelerate dialysis access graft thrombosis is based on the work of Himmelfarb and colleagues. In their trial aspirin appeared to increase the relative risk (RR=1.99) of graft thrombosis. They subsequently demonstrated that, in vitro, aspirin enhanced platelet-derived growth factor-induced vascular smooth muscle proliferation. Adding clopidogrel to aspirin in hemodialysis patients was associated with a significantly increased risk of bleeding and probably would not result in a reduced frequency of graft thrombosis. Although data concerning aspirin for primary or secondary prevention of cardiovascular disease in ESRD patients is not sufficient its efficacy is well proven in the general population. Currently, it seems not ethical to perform a randomized placebo controlled trial to evaluate the antiplatelet protective effect in these patients. The purpose of this study is to perform a prospective evaluation regarding the relationship between platelets function and cardiovascular events in patients with ESRD.

Methods The study will include 100-200 patients with ESRD, age 18 years or older, treated in the nephrology division of Assaf Harofeh medical center. Patients will be excluded if their platelets count will be lower then 50,000 cu/mm, if they have known hematologic malignancies, other solid malignancy with life expectancy of less then 1 year or if they are treated with Warfarin (Comadin). Patients will sign a written informed consent before their inclusion in the study.

The primary end points of the study are cardiovascular events including acute myocardial infarction (defined as symptoms + acute elevation of TnI), need for coronary artery disease revascularization, or acute cerebrovascular event (TIA or CVA) and mortality. The secondary end points are any hospitalization due to acute coronary syndrome, active bleeding with the need for blood transfusion and dialysis access graft thrombosis (time to thrombosis).

At the beginning of the study, blood will be taken for complete blood count including platelets count and mean platelets volume, serum electrolytes, albumin, blood lipids, Kt/V, troponin and two 5 ml aliquots from each blood collection will be separated and stored at -70co until analyzed for oxidative stress, homocysteine and highly sensitive CRP will be performed. Five mL of blood will be sent for platelets function assessment (described below).

The follow up period will be up to 2 years. During the follow up period, treatment with aspirin or clopidogrel will be given as needed and platelet function will be assessed after any change in the antiplatelets therapy. Patients who are being treated with aspirin, will continue to take the medication with no dose change unless they will have acute cardiovascular event or active bleeding. Patients will be treated with antihypertensive therapy, erythropoietin, calcium, vitamin D and other medications as needed.

Platelet Function Tests Cone-and-Platelet Analyzer This technology has been described elsewhere (40). Briefly, 200 µL of citrated blood was placed in a polystyrene well and subjected to a shear rate of 1300 sec-1 using a rotating conical disk for 2 minutes. The well was washed and stained by May-Gruenwald stain. Platelet adhesion was evaluated as the percentage of total area covered with platelets designated as surface coverage (%) and aggregation as the mean size of the surface-bound aggregates designated as average size (µ'm2) by use of an image analysis system (Galai).

Aspirin Response Assay 3.6µl Arachidonic Acid and 0.2ml blood will be added into a micro tube (2ml), (final Arachidonic Acid concentration 0.275 mM). The tube will be rotated on the tube mixer at 10rpm for 1 minute. 130µl will be placed in a well and tested with the cone and platelet analyzer.

Clopidogrel Response Assay 5µl ADP and 0.2ml blood will be added into a micro tube (2ml) (final ADP concentration 1.25µM). The tube will be rotated on the tube mixer at 10rpm for 1 minute. 130µl will be placed in a well and tested with the cone and platelet analyzer.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with end stage renal disease, age 18 years or older, treated in the nephrology division of Assaf Harofeh medical center.

Exclusion Criteria:

* Patients will be excluded if their platelets count will be lower then 50,000 cu/mm, if they have known hematologic malignancies, other solid malignancy with life expectancy of less then 1 year or if they are treated with Warfarin (Comadin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-09; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Study Chair — Assaf-Harofeh Medical Center; Mark Katz, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Nephrology Division, Aassaf-Harofeh Medical Center, Ẕerifin, Israel